CLINICAL TRIAL: NCT00582985
Title: An Open Label Phase 1 Dose Finding Study of TRC105 in Patients With Advanced or Metastatic Solid Cancer for Whom Curative Therapy is Unavailable
Brief Title: Open Label Phase 1 Dose Finding Study of TRC105 in Patients With Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Bryan Leigh, MD, Medical Monitor, TRACON Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105ST101
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Cancer; Neoplasm Metastasis
Keywords: Tracon; CD105; Anti CD105; TRC105; Phase 1; Cancer; Monoclonal antibody; Solid Tumor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TRC105 chimeric anti-CD105 antibody — TRC105 is a human/murine chimeric IgG1 antibody administered i.v. every two weeks (on days 1 and 15) or weekly (on days 1, 8, 15 and 22) of each 28 day cycle; until progression or unacceptable toxicity develops.

SUMMARY:
This study is being performed to evaluate the safety and tolerability of the TRC105 monoclonal antibody.

DETAILED DESCRIPTION:
In addition to safety, this study will also evaluate pharmacokinetics, tumor response and anti-TRC105 antibody formation.

ELIGIBILITY:
Inclusion Criteria:

* The patient has given informed consent.
* The patient is willing and able to abide by the protocol.
* The patient has cancer and curative therapy is unavailable.
* The patient is at least 18 years old.
* The patient has adequate ability to perform activities of daily living.
* Significant toxicities from prior therapy must have recovered.
* The patient has adequate organ function as assessed by laboratory test.

Exclusion Criteria:

* The patient weighs more than 264 lbs.
* The patient has a known allergy to gentamicin
* The patient has had prior treatment with high-dose chemotherapy requiring stem cell rescue
* The patient is currently on treatment on another therapeutic clinical trial or has received an investigational agent within 4 weeks prior to first dose with study drug
* The patient has had prior surgery (including open biopsy), radiation therapy or systemic therapy within 4 weeks of starting the study treatment
* The patient has hypertension > 160/90
* The patient has a history of CNS cancer
* The patient has an unstable medical condition including, but not limited to, cardiac disease, history of stroke, active hepatitis, or significant pericardial, pleural or peritoneal effusion
* The patient received recent thrombolytic or anticoagulant therapy
* The patient has lung cancer with central chest lesions
* The patient has had hemorrhage or unhealed wounds within 30 days of dosing
* The patient has used systemic corticosteroids within 3 months of dosing
* The patient has known HIV/AIDS
* The patient has a history of hypersensitivity reaction to human or mouse antibody products
* The patient is pregnant or breastfeeding.
* The patient has a history of peptic ulcer disease or gastritis within 6 months of dosing, unless complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 30 days of dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability will be evaluated | Through last patient last visit
Dose Limiting Toxicities | 28 day evaluation period

SECONDARY OUTCOMES:
Pharmacokinetics of TRC105 monoclonal antibody | through last patient last visit
Number of responses by tumor type | through last patient last visit

CONTACTS AND LOCATIONS:
Overall Officials: Bryan R Leigh, MD, Study Director — Tracon Pharmaceuticals Inc.
Locations (4):
- United States (4):
  - Scottsdale, Arizona
  - Santa Monica, California
  - Buffalo, New York
  - Durham, North Carolina

REFERENCES:
- [Derived] Seon BK, Haba A, Matsuno F, Takahashi N, Tsujie M, She X, Harada N, Uneda S, Tsujie T, Toi H, Tsai H, Haruta Y. Endoglin-targeted cancer therapy. Curr Drug Deliv. 2011 Jan;8(1):135-43. doi: 10.2174/156720111793663570. PMID 21034418